CLINICAL TRIAL: NCT05691257
Title: Study of the Safety and Efficacy of Roxadustat in the Treatment of Heart Failure With Chronic Kidney Disease and Anemia
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Jingyi Ren, Professor, China-Japan Friendship Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JRen
Record Dates: First submitted 2022-12-28; First posted 2023-01-19 (Actual); Last update posted 2023-01-20 (Actual); Status verified 2023-01

CONDITIONS: Heart Failure; Chronic Kidney Diseases; Anemia
Keywords: Roxadustat; Anemia; Biomarkers
MeSH Terms: conditions — Heart Failure; Renal Insufficiency, Chronic; Anemia | interventions — roxadustat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Roxadustat group (Experimental): Roxadustat group: patients with heart failure and chronic kidney disease and anemia treated with roxadustat and other anemia correction drugs.
  Interventions: Drug: Roxadustat; Drug: Recombinant human eythropoietin and/or Iron agents
- Control group (Other): Control group: patients with heart failure and chronic kidney disease and anemia who were treated with other drugs include: Recombinant human eythropoietin (RH-EPO), iron agents (ferrous succinate, polysaccharide iron complex, iron sucrose, etc.)
  Interventions: Drug: Recombinant human eythropoietin and/or Iron agents

INTERVENTIONS:
Drug: Roxadustat — The initial dose of roxadustat was given according to body weight, which was more than 60kg: 100mg (three times a week); Weight less than 60kg: 70mg (three times a week); 2 weeks later, the corresponding indexes were rechecked and medication was adjusted according to hemoglobin. The target is hemoglobin 100-120g/L.
  Reference for medication Method: The use of roxadustat is the same as the RCT study of roxadustat in the treatment of anemia and the drug instructions of roxadustat published by N Engl J Med in 2019.
  Arms: Roxadustat group
Drug: Recombinant human eythropoietin and/or Iron agents — Other drugs to treat anemia include: Recombinant human eythropoietin (RH-EPO), iron agents (ferrous succinate, polysaccharide iron complex, iron sucrose, etc.)

SUMMARY:
The purpose of this study is to conduct a a cohort study to evaluate the efficacy and safety of the efficacy and safety of roxadustat for the treatment of anemia, quality of life and cardiac function in patients with heart failure and chronic kidney disease.

DETAILED DESCRIPTION:
This is a cohort study in patients with anemia with heart failure complicated with chronic kidney disease, evaluating the the efficacy and safety of roxadustat. Patients were divided into roxadustat group and control group according to whether roxadustat was used or not. The efficacy and safety of roxadustat for the treatment of anemia, quality of life and cardiac function in patients with heart failure and chronic kidney disease will be evaluated.

The primary and secondary endpoints will be examined in subgroups determined by baseline variables reflecting demography, heart failure characteristics, diabetes status, kidney function, cardiac function, natriuretic peptide, dialysis, and additional co-morbidities, concomitant medications, and others.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, aged ≥18 years at the time of consent
2. Weight between 45-160kg
3. Definite diagnosis of heart failure: according to the diagnostic criteria for heart failure in "Chinese Heart Failure Diagnosis and Treatment Guidelines 2018"
4. eGFR <60mL/min/1.73 m^2 by CKD-EPI.
5. Diagnosed anemia: male hemoglobin <130 g/L, non-pregnant female hemoglobin <120 g/L.
6. Provision of signed informed consent prior to any study specific procedures.

Exclusion Criteria:

1. Acute or chronic active bleeding 6 months before enrollment.
2. Anemias due to thalassemia, sickle cell anemia, pure red aplastic anemia, hemolytic anemia, ect.
3. Thromboembolism requiring anticoagulation.
4. Severe Infection.
5. Hepatic impairment aspartate transaminase [AST] or alanine transaminase [ALT] >3x the upper limit of normal [ULN]; or total bilirubin >2x ULN at time of enrolment).
6. Severe malnutrition.
7. Women of child-bearing potential who are not willing to use a medically accepted method of contraception that is considered reliable in the judgment of the investigator OR women who have a positive pregnancy test at enrolment or randomization OR women who are breast-feeding.
8. Patients who have received roxadustat treatment or are allergic to roxadustat.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-02-01 (Estimated); Primary Completion 2023-08-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in the hemoglobin from baseline | up to 8 week
  Hemoglobin is calculated by the routine blood test

SECONDARY OUTCOMES:
Change in N-terminal Pro-brain Natriuretic Peptide (NT-proBNP) | Up to 8 weeks
  Change from baseline to week 12 in N-terminal pro-brain natriuretic peptide (NT-proBNP). Baseline value was defined as the mean of all available measurements from the screening visit until start of treatment with randomised study medication.
Change in Left Ventricular Systolic Function | Up to 24 weeks
  Change in left ventricular ejection fraction is assessed by two-dimensional directed M-mode echocardiography
Change in Left Ventricular End-Diastolic Diameter | Up to 24 weeks
  Change in left ventricular end-diastolic diameter is assessed by two-dimensional directed M-mode echocardiography
Change in Left Ventricular Diastolic Function | Up to 24 weeks
  Change in E/e' is assessed by two-dimensional directed M-mode echocardiography
Change in Low-density lipoprotein（LDL） | Up to 8 weeks
  Change from baseline to week 8 in Low-density lipoprotein（LDL）.Baseline value was defined as the mean of all available measurements from the screening visit until start of treatment with randomised study medication.
Change in Serum ferritin | Up to 8 weeks
  Change from baseline to week 8 in Serum ferritin.Baseline value was defined as the mean of all available measurements from the screening visit until start of treatment with randomised study medication.
Change in Transferrin saturation | Up to 8 weeks
  Change from baseline to week 8 in Transferrin saturation.Baseline value was defined as the mean of all available measurements from the screening visit until start of treatment with randomised study medication.
Change in Left atrial volume | Up to 24 weeks
  Change in left atrial volume is assessed by two-dimensional directed M-mode echocardiography
Change in Left atrial volume index | Up to 24 weeks
  Change in left atrial volume index is assessed by two-dimensional directed M-mode echocardiography

OTHER OUTCOMES:
Liver Injury | Up to 8 weeks
  Liver injury is defined as: i) a rise of alanine aminotransferase (ALT) or aspartate aminotransferase (AST) to 3 times above the upper limit of normal [ULN], or ii) a rise of total bilirubin to 2 times above the upper limit of normal [ULN]
Hyperkalemia | Up to 8 weeks
  Hyperkalemia is defined as：Serum potassium > 5.5 mmol/L
Thromboembolism | Up to 1 year
  Thromboembolism is defined as：Deep vein thrombosis at follow-up

IPD SHARING:
Plan to Share IPD: Undecided